CLINICAL TRIAL: NCT00298649
Title: Reducing Farmworkers Exposure to Agricultural Chemicals
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 8739-CP-001
Record Dates: First submitted 2006-03-01; First posted 2006-03-02 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2006-03

CONDITIONS: Pesticide Safety
Keywords: pesticide safety; migrant and seasonal farmworkers; Latino/Hispanic; agricultural health; occupational health

INTERVENTIONS:
Behavioral: Lay Health Advisor

SUMMARY:
The goal of this project is to develop and test the effectiveness of a Lay Health Advisor program to teach migrant and seasonal farmworkers about pesticide safety in their homes. This is a community-based collaborative research project in which we first conduct in-depth interviews with farmworkers to learn about their knowledge and beliefs relative to pesticide exposure in the home, and, second, develop the content of the Lay Health Advisor program based on this formative information. We will evaluate this program by conducting pre- and post-test interviews with farmworkers, and comparing safety and knowledge to a control group who receive other important health education.

DETAILED DESCRIPTION:
?La Familia! extends collaboration between the North Carolina Farmworkers' Project (NCFP), a grassroots community based organization, and environmental health researchers at Wake Forest University School of Medicine to evaluate a Lay Health Advisor (LHA) model to reduce pesticide exposure among farmworker families. The proposed research builds on PACE, Preventing Agricultural Chemical Exposure among North Carolina Farmworkers (R21 ES08739), a highly successful workplace intervention to reduce migrant and seasonal farmworker pesticide exposure. With ?La Familia!, the PACE focus shifts to exposure of farmworker families, particularly children, and expands work with the North Carolina farmworker community to workers in the western region of the state. ?La Familia!'s specific aims are to: (1) document and assess farmworker knowledge, beliefs and perceptions of pesticide exposure of all family members, particularly as they relate to exposure of children; (2) identify pathways for environmental exposure of farmworker children to pesticides; (3) develop, implement, and evaluate a culturally appropriate LHA intervention to reduce pesticide exposure of children (aged 18-48 mo) in farmworker homes; and (4) compile and disseminate the final intervention program to other farmworker communities and farmworker service providers. A model of community participation will be implemented throughout the 5 project years. Formative research (in-depth interviews; pathway exposure assessment) will be completed in Years 1 and 2. Using the formative results in a PRECEDE-PROCEED framework, the content and format of the LHA intervention will be developed in Year 2. This intervention (and a revision) will be evaluated in Years 3 and 4 using a group randomized design. End-points will include change in knowledge of pesticide exposure routes for children and ways to reduce their exposure; change in exposure-related behaviors; and changes in household dust levels. In the final year, support will continue for the LHA program as part of the process of NCFP developing its health outreach mission in western NC., while the results of the project are disseminated to regional and national farmworker groups, to those providing health care to farmworkers, and in the research literature.

ELIGIBILITY:
Inclusion Criteria

* Adults
* At least household resident employed in farmwork
* At least one coresident child

Exclusion Criteria

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2002-07; Study Completion 2004-10

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A. Arcury, Ph.D., Principal Investigator — Department of Family and Community Medicine, Wake Forest University School of Medicine
Locations (1):
- Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States

REFERENCES:
- [Result] Arcury TA, Quandt SA. Pesticides at work and at home: exposure of migrant farmworkers. Lancet. 2003 Dec 13;362(9400):2021. doi: 10.1016/S0140-6736(03)15027-1. No abstract available. PMID 14686376
- [Result] Quandt SA, Arcury TA, Rao P, Snively BM, Camann DE, Doran AM, Yau AY, Hoppin JA, Jackson DS. Agricultural and residential pesticides in wipe samples from farmworker family residences in North Carolina and Virginia. Environ Health Perspect. 2004 Mar;112(3):382-7. doi: 10.1289/ehp.6554. PMID 14998757
- [Result] Quandt SA, Doran AM, Rao P, Hoppin JA, Snively BM, Arcury TA. Reporting pesticide assessment results to farmworker families: development, implementation, and evaluation of a risk communication strategy. Environ Health Perspect. 2004 Apr;112(5):636-42. doi: 10.1289/ehp.6754. PMID 15064174
- [Result] Quandt SA, Arcury TA, Mellen, BG, Rao P, Camann DE, Coran AM, Yau A, Hoppin JA, Jackson DS. Pesticides in wipes from farmworker residences in North Carolina. In Proceedings of Indoor Air 2002, H. Levin, ed., Santa Cruz, CA, Vol. 4:900-905, 2002.
- [Result] Rao P, Arcury TA, Quandt SA, Doran A. North Carolina Growers' and Extension Agents' Perceptions of Latino Farmworker Pesticide Exposure. Hum Organ. 2004 Summer;63(2):151-161. doi: 10.17730/humo.63.2.qdyhan8n1ngkf2rk. PMID 31579320
- [Result] Arcury TA, Quandt SA, Rao P, Doran AM, Snively BM, Barr DB, Hoppin JA, Davis SW. Organophosphate Pesticide Exposure in Farmworker Family Members in Western North Carolina and Virginia: Case Comparisons. Hum Organ. 2005 Spring;64(1):40-51. PMID 31467451
- [Result] Rao P, Quandt SA, Doran AM, Snively BM, Arcury TA. Pesticides in the homes of farmworkers: Latino mothers' perceptions of risk to their children's health. Health Educ Behav. 2007 Apr;34(2):335-53. doi: 10.1177/1090198106288045. Epub 2006 May 31. PMID 16740507
- [Result] Early J, Davis SW, Quandt SA, Rao P, Snively BM, Arcury TA. Housing characteristics of farmworker families in North Carolina. J Immigr Minor Health. 2006 Apr;8(2):173-84. doi: 10.1007/s10903-006-8525-1. PMID 16649132
- [Result] Rao P, Gentry AL, Quandt SA, Davis SW, Snively BM, Arcury TA. Pesticide safety behaviors in Latino farmworker family households. Am J Ind Med. 2006 Apr;49(4):271-80. doi: 10.1002/ajim.20277. PMID 16550565